CLINICAL TRIAL: NCT00141271
Title: A Six-Week, Randomized, Double-Blind, Multicenter, Fixed-Flexible Dose, Placebo-Controlled Study Evaluating the Efficacy and Safety of Oral Ziprasidone in Outpatients With Bipolar I Depression
Brief Title: A Six-Week Study Evaluating The Efficacy And Safety Of Geodon In Patients With A Diagnosis Of Bipolar I Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1281136
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Results first posted 2009-03-24 (Estimated); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Bipolar Disorder
Keywords: Bipolar I Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — ziprasidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 20-40mg BID arm (Active Comparator)
  Interventions: Drug: Geodon (Ziprasidone)
- 60-80mg bid arm (Active Comparator)
  Interventions: Drug: Geodon (Ziprasidone)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Geodon (Ziprasidone) — Subjects will start at 20mg bid days 1-6, then flexible dosing starting on day 7 between 20-40mg bid (20mg bid or 40mg bid) for the remainder of the 6 week trial
  Arms: 20-40mg BID arm
Drug: Geodon (Ziprasidone) — Subjects will start at 20mg bid days 1-2, then 40mg bid days 3-4, them 60mg bid for days 5-6 then flexible dosing starting on day 7 between 60-80mg bid (60 mg bid or 80mg bid) for the remainder of the 6 week trial
  Arms: 60-80mg bid arm
Drug: Placebo — Subjects will start on placebo and remain on placebo for the remainder of the 6 week trial
  Arms: Placebo

SUMMARY:
This is a 6-week trial that evaluates the efficacy and safety of Geodon (ziprasidone) in outpatient subjects ages 18 and older with Bipolar Disorder type I, depressed. Subjects are required to undergo a washout period of at least 7 days of any prior med.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a primary diagnosis of Bipolar I Disorder, most recent episode depressed, with or without rapid cycling, without psychotic features, as defined in Diagnostic and Statistical Manual (of Mental Disorders) - Fourth Edition - Text Revision (DSM-IV-TR) (296.5X) and confirmed by a structured Mini International Neuropsychiatric Interview (MINI)

Exclusion Criteria:

* Subjects with a DSM-IV TR diagnosis of schizophrenia (295.XX), schizoaffective disorder (295.70), schizophreniform disorder (295.40), delusional disorder (297.1), or psychotic disorder not otherwise specified (298.9).
* Subjects with other DSM-IV TR Axis I or Axis II disorder (in addition to Bipolar I disorder) are ineligible if the comorbid condition is clinically unstable, requires treatment, or has been a primary focus of treatment within the 6 month period prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Actual)
Dates: Start 2005-07; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (63):
- United States (63):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Dana Point, California
  - Pfizer Investigational Site, La Mesa, California
  - Pfizer Investigational Site, Laguna Hills, California
  - Pfizer Investigational Site, Oceanside, California
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Santa Ana, California
  - Pfizer Investigational Site, Torrance, California
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Hialeah, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, North Miami, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Winter Park, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Maywood, Illinois
  - Pfizer Investigational Site, Naperville, Illinois
  - Pfizer Investigational Site, Schaumburg, Illinois
  - Pfizer Investigational Site, Greenwood, Indiana
  - Pfizer Investigational Site, Lafayette, Indiana
  - Pfizer Investigational Site, Prarie Village, Kansas
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Flowood, Mississippi
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Clementon, New Jersey
  - Pfizer Investigational Site, Toms River, New Jersey
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Staten Island, New York
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Mayfield, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Columbia, South Carolina
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Bellaire, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, DeSoto, Texas
  - Pfizer Investigational Site, Galveston, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Irving, Texas
  - Pfizer Investigational Site, Plano, Texas
  - Pfizer Investigational Site, Richardson, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Wichita Falls, Texas
  - Pfizer Investigational Site, Arlington, Virginia
  - Pfizer Investigational Site, Falls Church, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Virginia Beach, Virginia
  - Pfizer Investigational Site, Kirkland, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin
  - Pfizer Investigational Site, West Allis, Wisconsin

REFERENCES:
- [Derived] Keefe RS, Fox KH, Davis VG, Kennel C, Walker TM, Burdick KE, Harvey PD. The Brief Assessment of Cognition In Affective Disorders (BAC-A):performance of patients with bipolar depression and healthy controls. J Affect Disord. 2014 Sep;166:86-92. doi: 10.1016/j.jad.2014.05.002. Epub 2014 May 11. PMID 25012414
- [Derived] Gao K, Pappadopulos E, Karayal ON, Kolluri S, Calabrese JR. Risk for adverse events and discontinuation due to adverse events of ziprasidone monotherapy relative to placebo in the acute treatment of bipolar depression, mania, and schizophrenia. J Clin Psychopharmacol. 2013 Jun;33(3):425-31. doi: 10.1097/JCP.0b013e3182917f3f. PMID 23609405
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281136&StudyName=A%20Six-Week%20Study%20Evaluating%20The%20Efficacy%20And%20Safety%20Of%20Geodon%20In%20Patients%20With%20A%20Diagnosis%20Of%20Bipolar%20I%20Depression

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 56 centers in the US
Pre-assignment Details: 7-day washout:psychotropic drugs & lithium. 4-week washout: monoamine oxidase inhibitors, fluoxetine alone or in combination with olanzapine. Depot neuroleptic Discontinued (DC'd) 6 mo prior to entry. 536 subjects enrolled: 504 assigned to drug; 32 not assigned:18 lost to follow up, 5 DC'd study, 9 didn't take/receive study drug for other reasons.
Groups:
- 120-160mg Ziprasidone: Subjects were assigned to a ziprasidone fixed-flexible dosing arm: 60-80 milligram (mg) BID (twice a day)
- 40-80 mg Ziprasidone: Subjects were assigned to a ziprasidone fixed-flexible dosing arm: 20-40 milligram (mg) twice a day (BID)
- Placebo: Subjects were assigned to placebo
Period: Overall Study
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Started | 171 | 165 | 168
Completed | 91 | 102 | 111
Not Completed | 80 | 63 | 57
Not completed — Adverse Event | 31 | 19 | 17
Not completed — Laboratory Abnormality | 2 | 1 | 1
Not completed — Lack of Efficacy | 7 | 7 | 3
Not completed — Lost to Follow-up | 15 | 15 | 21
Not completed — Withdrawal by Subject | 14 | 9 | 10
Not completed — Other | 11 | 12 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo | Total
Number analyzed (Participants) | 171 | 165 | 168 | 504
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (12.9) | 40.0 (11.4) | 39.3 (11.2) | 39.9 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 101 | 92 | 284
  Male | 80 | 64 | 76 | 220

OUTCOME MEASURES:

1. Primary Outcome: Change in Montgomery-Asberg Depression Rating Scale (MADRS)Total Score
Description: Change is observed value at each visit minus baseline value. Overall is average response of Weeks 1 - 6. MADRS is 10-item instrument measuring depression; scale 0(Normal) and 6(most abnormal). Total possible score is 0 - 60.
Time Frame: Baseline to 6 weeks
Population: Intent to treat (ITT) population observed cases
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
score on scale
  Week 1 (n=161, 153, 159) | -6.07 (0.62) | -7.66 (0.73) | -5.75 (0.65)
  Week 2 (n=135, 142, 146) | -10.12 (0.79) | -10.20 (0.82) | -9.47 (0.77)
  Week 3 (n=120, 131, 138) | -11.61 (0.88) | -12.93 (0.85) | -11.37 (0.81)
  Week 4 (n=106, 126, 131) | -12.54 (0.88) | -13.87 (0.91) | -12.49 (0.82)
  Week 5 (n=99, 115, 123) | -14.25 (0.94) | -14.53 (0.90) | -12.99 (0.97)
  Week 6 (n=95, 107, 115) | -13.81 (1.02) | -14.77 (0.97) | -13.25 (1.00)
  Overall (n=166, 158, 162) | -11.40 (0.73) | -12.33 (0.74) | -10.89 (0.72)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Week 1; Test type: Superiority or Other; p = 0.6409, Mixed Models Analysis — Hochberg's adjustment was used for multiple comparisons adjustment; Fixed categorical: treatment, rapid cycling, center, visit, prior hosp & treatment-by-visit interaction & fixed continuous effect of baseline value
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 1; Test type: Superiority or Other; p = 0.0140, Mixed Models Analysis — Hochberg's adjustment used for multiple comparisons adjustment; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: 120-160mg Ziprasidone vs Placebo; Week 2; Test type: Superiority or Other; p = 0.4840, Mixed Models Analysis — Hochberg's adjustment used for multiple comparisons adjustment; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 2; Test type: Superiority or Other; p = 0.4444, Mixed Models Analysis — Hochberg's adjustment used for multiple comparisons adjustment; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: 120-160mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.8129, Mixed Models Analysis — Hochberg's adjustment used for multiple comparisons adjustment; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.1105, Mixed Models Analysis — Hochberg's adjustment used for multiple comparisons adjustment; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: 120-160mg Ziprasidone vs Placebo; Week 4; Test type: Superiority or Other; p = 0.9582, Mixed Models Analysis — Hochberg's adjustment used for multiple comparisons adjustment; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 4; Test type: Superiority or Other; p = 0.1893, Mixed Models Analysis — Hochberg's adjustment used for multiple comparisons adjustment; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: 120-160mg Ziprasidone vs Placebo; Week 5; Test type: Superiority or Other; p = 0.2924, Mixed Models Analysis — Hochberg's adjustment used for multiple comparisons adjustment; Hochberg's adjustment used for multiple comparisons adjustment
Statistical Analysis 10: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 5; Test type: Superiority or Other; p = 0.1897, Mixed Models Analysis — Hochberg's adjustment used for multiple comparisons adjustment; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: 120-160mg Ziprasidone vs Placebo; Week 6 An estimated sample size of 180 was needed per treatment arm in order to achieve 85% power to detect a treatment difference of 3.5 in the mean change from baseline to Week 6 in MADRS total score with a two-sided t-test at the 0.05 significance level. The common standard deviation was estimated as 11.0. The null hypotheses for the primary parameter is equality of mean change from baseline to Week 6 in MADRS total score between ziprasidone and placebo groups; Test type: Superiority or Other; p = 0.6608, Mixed Models Analysis — Hochberg's adjustment used for multiple comparisons adjustment; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: 40-80 mg Ziprasidone vs Placebo; [analysis description as in outcome 1, analysis 11]; Test type: Superiority or Other; p = 0.2148, Mixed Models Analysis — Hochberg's adjustment used for multiple comparisons adjustment; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: 120-160mg Ziprasidone vs Placebo; Overall; Test type: Superiority or Other; p = 0.5290, Mixed Models Analysis — Hochberg's adjustment used for multiple comparisons adjustment; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: 40-80 mg Ziprasidone vs Placebo; Overall; Test type: Superiority or Other; p = 0.0811, Mixed Models Analysis — Hochberg's adjustment used for multiple comparisons adjustment; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Response Greater Than or Equal to 50 Percent Decrease From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS)Total Score
Description: Participants with MADRS Total Score greater or equal to 50 percent decrease from baseline responded yes; others responded no. Endpoint is last observation carried forward (LOCF) among Week 1 - Week 6; MADRS is 10-item instrument measuring depression; scale range 0(Normal) and 6 (most abnormal). Total possible score is 0 - 60
Time Frame: Baseline to 6 weeks
Population: Intent to treat (ITT) population observed cases.
  Not all subjects answered at each Week
Measure: Number; unit: Participants
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
Participants
  Week 1: Yes | 19 | 32 | 26
  Week 1: No | 142 | 121 | 133
  Week 2 : Yes | 51 | 50 | 51
  Week 2: No | 84 | 92 | 95
  Week 3: Yes | 57 | 67 | 60
  Week 3: No | 63 | 64 | 78
  Week 4: Yes | 56 | 70 | 68
  Week 4: No | 50 | 56 | 63
  Week 5: Yes | 67 | 74 | 71
  Week 5: No | 32 | 41 | 52
  Week 6: Yes | 58 | 69 | 67
  Week 6: No | 37 | 38 | 48
  Endpoint: Yes | 76 | 83 | 80
  Endpoint: No | 90 | 75 | 82
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Week 1; Test type: Superiority or Other; p = 0.2287, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; CMH test stratified by study center and rapid cycling strata was used to compare remission and response rates between ziprasidone and placebo groups
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Week1; Test type: Superiority or Other; p = 0.4734, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: 120-160mg Ziprasidone vs Placebo; Week 2; Test type: Superiority or Other; p = 0.7401, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 2; Test type: Superiority or Other; p = 0.7904, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: 120-160mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.5274, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.1059, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: 120-160mg Ziprasidone vs Placebo; Week 4; Test type: Superiority or Other; p = 0.8871, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 4; Test type: Superiority or Other; p = 0.6939, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: 120-160mg Ziprasidone vs Placebo; Week 5; Test type: Superiority or Other; p = 0.1044, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 5; Test type: Superiority or Other; p = 0.3132, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: 120-160mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.6978, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.3228, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.6432, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 14: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.5989, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]

3. Secondary Outcome: Response Greater Than or Equal to 50 Percent Decrease From Baseline in Hamilton Depression Rating Scale (HAM-D 17) Total Score
Description: Participants with greater than or equal to 50 percent decrease from baseline in HAMD-17 total score responded yes; others responded no. Endpoint is LOCF endpoint among Week 1 - 6; Total score is first 17 items of HAM-D 25: measures range of depressive symptoms; scale 0-2 or 0-4 with higher scores being more severe. Total possible score 0 - 52.
Time Frame: Baseline to 6 weeks
Population: Intent to treat (ITT) population observed cases. Endpoint is LOCF endpoint among Week 1 through Week 6
  Not all subjects answered each Week.
Measure: Number; unit: participants
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
participants
  Week 3: Yes | 60 | 67 | 61
  Week 3: No | 87 | 82 | 87
  Week 6: Yes | 64 | 73 | 73
  Week 6: No | 40 | 44 | 52
  Endpoint: Yes | 74 | 82 | 81
  Endpoint: No | 77 | 68 | 72
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.8921, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.4350, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: 120-160mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.5620, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.6959, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.7865, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.7564, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]

4. Secondary Outcome: Change in Global Assessment of Functioning (GAF)at Endpoint, Last Observation Carried Forward (LOCF)
Description: Change is observed value at endpoint minus baseline value. Endpoint is Last Observation Carried Forward (LOCF) endpoint among Week 1 - 6; GAF is used to assess global psychological, social, & occupational functioning; 100=normal and 0=greatest abnormality
Time Frame: Baseline, 6 Weeks LOCF
Population: Intent to treat (ITT) population observed cases, Last Observation Carried Forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
score on scale | 10.11 (1.38) | 11.72 (1.37) | 11.19 (1.40)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.4327, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; Model included model terms of treatment, rapid cycling, center, prior hospitalization status, as well as baseline value as a covariate
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.7041, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 4, analysis 1]

5. Secondary Outcome: Remission as Measured by Montgomery-Asberg Depression Rating Scale (MADRS) Total Score Less Than or Equal to 12
Description: Response was Yes if MADRS Total Score was less than, equal to 12, if not, response was no. Endpoint is LOCF endpoint among Week 1 through 6; MADRS is 10-item instrument measuring depression; scale range 0(Normal) and 6(most abnormal)
Time Frame: Baseline to 6 weeks
Population: ITT Observed Cases.Endpoint is LOCF endpoint among Week 1 through Week 6;
  Not all subjects answered each week.
Measure: Number; unit: participants
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
participants
  Week 1; Yes | 18 | 27 | 25
  Week 1; No | 143 | 126 | 134
  Week 2; Yes | 48 | 41 | 44
  Week 2; No | 87 | 101 | 102
  Week 3; Yes | 56 | 61 | 55
  Week 3; No | 64 | 70 | 83
  Week 4; Yes | 55 | 65 | 66
  Week 4; No | 51 | 61 | 65
  Week 5; Yes | 65 | 66 | 66
  Week 5; No | 34 | 49 | 57
  Week 6; Yes | 58 | 63 | 61
  Week 6; No | 37 | 44 | 54
  Endpoint; Yes | 73 | 72 | 73
  Endpoint; No | 93 | 86 | 89
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Week 1; Test type: Superiority or Other; p = 0.2076, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 1; Test type: Superiority or Other; p = 0.7449, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: 120-160mg Ziprasidone vs Placebo; Week 2; Test type: Superiority or Other; p = 0.4399, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 2; Test type: Superiority or Other; p = 0.7107, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: 120-160mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.4765, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.2564, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: 120-160mg Ziprasidone vs Placebo; Week 4; Test type: Superiority or Other; p = 0.8063, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 4; Test type: Superiority or Other; p = 0.9855, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: 120-160mg Ziprasidone vs Placebo; Week 5; Test type: Superiority or Other; p = 0.0599, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 5; Test type: Superiority or Other; p = 0.7364, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: 120-160mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.3048, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.5139, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.9356, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 14: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.9428, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]

6. Secondary Outcome: Remission as Measured by Hamilton Depression (HAM-D 17) Total Score Less Than or Equal to 7
Description: Response was yes when HAM-D 17 total score was less than or equal to 7 , if not, response was no. Endpoint is LOCF endpoint among Week 1 through Week 6. Total score is first 17 items of the HAM-D 25,which measures the range of depressive symptoms; scale 0-2 or 0-4 with higher scores being more severe. Total possible score 0 - 52.
Time Frame: Baseline to 6 weeks
Population: ITT Observed Cases.Endpoint is LOCF endpoint among Week 1 through Week 6
  Not all subjects answered each week.
Measure: Number; unit: Participants
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
Participants
  Week 3; Yes | 27 | 30 | 35
  Week 3; No | 120 | 119 | 113
  Week 6; Yes | 41 | 43 | 43
  Week 6; No | 63 | 74 | 82
  Endpoint: Yes | 45 | 44 | 47
  Endpoint: No | 106 | 106 | 106
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.3888, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.3122, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: 120-160mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.3323, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.8781, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.9485, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.7331, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]

7. Secondary Outcome: Change in Hamilton Depression (HAM-D 17) Total Score
Description: Change is observed value at each visit minus baseline value. Endpoint is LOCF endpoint among Week 1 through Week 6. Total score is first 17 items of the HAM-D 25, which measures the range of depressive symptoms patient currently experiencing; scale 0-2 or 0-4; 0=absent or not depressed, 2 or 4=most severe or extreme. Total possible score 0 - 52.
Time Frame: Baseline to 6 weeks
Population: ITT Population Observed Cases. Endpoint is LOCF endpoint among Week 1 through Week 6.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
score on scale
  Week 3 (n= 147, 149, 148) | -9.56 (0.82) | -10.58 (0.81) | -10.13 (0.82)
  Week 6 (n= 104,117,125) | -12.37 (1.12) | -12.82 (1.06) | -11.30 (1.06)
  Endpoint (n= 151,150,153) | -10.48 (0.95) | -11.48 (0.95) | -10.60 (0.95)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.4869, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.5813, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: 120-160mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.3303, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.1546, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.8982, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.3586, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]

8. Secondary Outcome: Change in Hamilton Anxiety Rating (HAM-A)
Description: Change is observed value at each visit minus baseline value. Endpoint is LOCF endpoint among Week 1 through Week 6. HAM-A is a 14-item scale: rates intensity of psychic anxiety and somatic anxiety on a 5-point severity scale (range: 0=not present to 4=very severe). Total possible score is 0 - 56.
Time Frame: Baseline to 6 weeks
Population: ITT population Observed Cases. Endpoint is LOCF endpoint among Week 1 through Week 6
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
score on scale
  Week 3 (n= 147, 148, 147) | -5.54 (0.74) | -6.46 (0.74) | -6.79 (0.74)
  Week 6 (n= 104, 117, 124) | -7.63 (0.94) | -7.46 (0.89) | -6.73 (0.89)
  Endpoint (n= 151, 150, 152) | -6.40 (0.81) | -6.75 (0.81) | -6.82 (0.82)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.0896, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.6534, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: 120-160mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.3270, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.4099, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.6104, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.9359, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]

9. Secondary Outcome: Change in Total Score of Young Mania Rating Scale (YMRS)
Description: Change is observed value at each visit minus baseline value. Overall is average response of Weeks 1 - 6. YMRS: 11 item instrument with scale 0 to 4 for 7 items and 0 to 8 for 4 items; 0=normal; 4 or 8=most abnormal. Total possible score is 0 - 60.
Time Frame: Baseline to 6 weeks
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
score on scale
  Week 1 (n = 140,131, 132) | 0.05 (0.34) | 0.64 (0.41) | -0.08 (0.33)
  Week 2 (n = 114,124,123) | 0.16 (0.38) | 0.64 (0.41) | 0.51 (0.37)
  Week 3 (n = 120, 130, 138) | -0.03 (0.44) | 0.11 (0.39) | 0.05 (0.40)
  Week 4 (n = 93, 116, 116) | -0.09 (0.43) | 0.19 (0.49) | -0.73 (0.41)
  Week 5 (n = 87, 105, 109) | -0.89 (0.43) | -0.82 (0.43) | -0.28 (0.45)
  Week 6 (n = 95, 107, 115) | -0.86 (0.42) | -0.03 (0.50) | -1.00 (0.42)
  Overall (n = 161, 158, 161) | -0.27 (0.33) | 0.12 (0.36) | -0.26 (0.32)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Week 1; Test type: Superiority or Other; p = 0.6924, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 1; Test type: Superiority or Other; p = 0.0800, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: 120-160mg Ziprasidone vs Placebo; Week 2; Test type: Superiority or Other; p = 0.4238, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 2; Test type: Superiority or Other; p = 0.7714, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: 120-160mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.8731, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.8926, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: 120-160mg Ziprasidone vs Placebo; Week 4; Test type: Superiority or Other; p = 0.2072, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 4; Test type: Superiority or Other; p = 0.1042, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: 120-160mg Ziprasidone vs Placebo; Week 5; Test type: Superiority or Other; p = 0.2695, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 5; Test type: Superiority or Other; p = 0.3245, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: 120-160mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.7791, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.0999, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: 120-160mg Ziprasidone vs Placebo; Overall; Test type: Superiority or Other; p = 0.9543, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: 40-80 mg Ziprasidone vs Placebo; Overall; Test type: Superiority or Other; p = 0.3153, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]

10. Secondary Outcome: Change in Assessment of Global Clinical Severity of Symptoms (CGI-S)
Description: Change is observed value at each visit minus baseline value. Overall is average response of Weeks 1 - 6. CGI-S measures severity of patient's mental illness. Scale range: 0 = not assessed, 1 = normal, 7 = among most extremely ill
Time Frame: Baseline to 6 weeks
Population: ITT population Observed Cases
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
score on scale
  Week 1 (n=161, 152, 158) | -0.05 (0.08) | -0.47 (0.07) | -0.42 (0.07)
  Week 2 (n=133, 142, 147) | -0.84 (0.09) | -0.82 (0.09) | -0.75 (0.09)
  Week 3 (n=119, 131, 137) | -0.90 (0.11) | -1.15 (0.10) | -0.93 (0.09)
  Week 4 (n=105, 126, 130) | -1.14 (0.11) | -1.23 (0.11) | -1.14 (0.10)
  Week 5 (n=98, 115, 123) | -1.33 (0.11) | -1.35 (0.12) | -1.23 (0.11)
  Week 6 (n=94, 107, 115) | -1.38 (0.12) | -1.38 (0.12) | -1.35 (0.12)
  Overall (n=165, 158, 162) | -1.02 (0.09) | -1.07 (0.09) | -0.97 (0.08)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Week 1; Test type: Superiority or Other; p = 0.2878, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 1; Test type: Superiority or Other; p = 0.4481, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: 120-160mg Ziprasidone vs Placebo; Week 2; Test type: Superiority or Other; p = 0.4099, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 2; Test type: Superiority or Other; p = 0.5093, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: 120-160mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.8048, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.0552, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: 120-160mg Ziprasidone vs Placebo; Week 4; Test type: Superiority or Other; p = 0.9795, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 4; Test type: Superiority or Other; p = 0.5073, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: 120-160mg Ziprasidone vs Placebo; Week 5; Test type: Superiority or Other; p = 0.4882, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 5; Test type: Superiority or Other; p = 0.3967, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: 120-160mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.8276, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.8502, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: 120-160mg Ziprasidone vs Placebo; Overall; Test type: Superiority or Other; p = 0.6343, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: 40-80 mg Ziprasidone vs Placebo; Overall; Test type: Superiority or Other; p = 0.3082, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]

11. Secondary Outcome: Change in Global Clinical Improvement of Symptoms (CGI -I)
Description: Change is observed value at each visit minus baseline value. Overall is average response of Weeks 1 - 6. CGI-I is an instrument for Global assessment of improvement in patient's condition. Scale range: 0=not assessed, 1=very much improved, 7=very much worse
Time Frame: Baseline to 6 weeks
Population: ITT population Observed Cases
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
score on scale
  Week 1 (n=162, 152, 158) | 3.34 (0.09) | 3.17 (0.09) | 3.38 (0.09)
  Week 2 (n=134, 142, 147) | 2.86 (0.11) | 2.82 (0.10) | 3.01 (0.10)
  Week 3 (n=120,131,137) | 2.90 (0.13) | 2.62 (0.11) | 2.83 (0.10)
  Week 4 (n=106,126,130) | 2.54 (0.11) | 2.53 (0.11) | 2.55 (0.10)
  Week 5 (n=99, 115, 123) | 2.47 (0.12) | 2.48 (0.12) | 2.59 (0.12)
  Week 6 (n=95,107, 115) | 2.49 (0.13) | 2.43 (0.13) | 2.52 (0.12)
  Overall (n=166, 158, 162) | 2.77 (0.10) | 2.67 (0.09) | 2.81 (0.09)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Week 1; Test type: Superiority or Other; p = 0.6932, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 1; Test type: Superiority or Other; p = 0.0287, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: 120-160mg Ziprasidone vs Placebo; Week 2; Test type: Superiority or Other; p = 0.2128, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 2; Test type: Superiority or Other; p = 0.1118, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: 120-160mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.6144, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.0899, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: 120-160mg Ziprasidone vs Placebo; Week 4; Test type: Superiority or Other; p = 0.8819, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 4; Test type: Superiority or Other; p = 0.8374, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: 120-160mg Ziprasidone vs Placebo; Week 5; Test type: Superiority or Other; p = 0.3925, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 5; Test type: Superiority or Other; p = 0.4182, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: 120-160mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.8586, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.5490, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: 120-160mg Ziprasidone vs Placebo; Overall; Test type: Superiority or Other; p = 0.6292, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: 40-80 mg Ziprasidone vs Placebo; Overall; Test type: Superiority or Other; p = 0.1473, Mixed Models Analysis — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 1, analysis 1]

12. Secondary Outcome: Change in Total Score in Hamilton Depression (HAM-D 25)
Description: Change: observed value at each visit minus baseline value. Endpoint is Last Observation Carried Forward (LOCF) endpoint among Week 1 through Week 6. HAM-D 25: measures the range of depressive symptoms experienced. 25 Items with Scale range:0-2 or 0-4; 0=absent or not depressed, 2 or 4=most severe or extreme.Total possible score is 0 - 72.
Time Frame: Baseline to 6 Weeks
Population: ITT Population Observed Cases. Endpoint is LOCF endpoint among Week 1 through Week 6.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
score on scale
  Week 3 (n= 147, 149, 147) | -11.02 (0.98) | -12.16 (0.97) | -12.25 (0.98)
  Week 6 (n= 104, 117, 125) | -14.59 (1.32) | -15.08 (1.25) | -13.74 (1.24)
  Endpoint (n= 151, 150, 153) | -12.25 (1.11) | -13.36 (1.11) | -12.78 (1.11)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.2058, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.9254, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: 120-160mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.5071, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.2858, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.6298, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.6034, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 4, analysis 1]

13. Secondary Outcome: Response as Measured by CGI-I Score Less Than or Equal to 2
Description: Response each week was yes if CGI-I score less than or equal to 2 (much or very much improved), if not, response was no; Endpoint is LOCF endpoint among Week 1 through Week 6. CGI-I is a Global assessment of improvement in patient's condition. Scale range: 0=not assessed, 1=very much improved, 7=very much worse
Time Frame: Week 1 through Week 6 (endpoint)
Population: ITT Population Observed cases. Endpoint is LOCF endpoint among Week 1 through Week 6.
  Not all subjects answered each week.
Measure: Number; unit: Participants
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
Participants
  Week 1; Yes | 20 | 34 | 28
  Week 1; No | 142 | 118 | 130
  Week 2; Yes | 52 | 54 | 50
  Week 2; No | 82 | 88 | 97
  Week 3; Yes | 51 | 71 | 58
  Week 3; No | 69 | 60 | 79
  Week 4; Yes | 68 | 76 | 70
  Week 4; No | 38 | 50 | 60
  Week 5; Yes | 69 | 74 | 73
  Week 5; No | 30 | 41 | 50
  Week 6; Yes | 60 | 76 | 66
  Week 6; No | 35 | 31 | 49
  Endpoint; Yes | 74 | 83 | 77
  Endpoint; No | 92 | 75 | 85
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Week 1; Test type: Superiority or Other; p = 0.1454, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 1; Test type: Superiority or Other; p = 0.2672, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: 120-160mg Ziprasidone vs Placebo; Week 2; Test type: Superiority or Other; p = 0.2614, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 2; Test type: Superiority or Other; p = 0.2143, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: 120-160mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.6997, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.0128, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: 120-160mg Ziprasidone vs Placebo; Week 4; Test type: Superiority or Other; p = 0.1144, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 4; Test type: Superiority or Other; p = 0.1483, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: 120-160mg Ziprasidone vs Placebo; Week 5; Test type: Superiority or Other; p = 0.0674, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 5; Test type: Superiority or Other; p = 0.2900, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: 120-160mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.5482, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.0303, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.6143, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 14: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.3385, Cochran-Mantel-Haenszel — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 2, analysis 1]

14. Secondary Outcome: Change in Sheehan Disability Scale (SDS) Total Score at Endpoint
Description: Observed value each visit minus baseline value. Endpoint is LOCF Week 1 through Week 6. SDS: patient rated measure of disability and impairment in 3 items: work/school, social life, family life/home responsibilities:0(no disruption)- 10(extreme disruption). Total possible is 30.
Time Frame: Baseline to Week 6
Population: ITT Population Observed cases. Endpoint is LOCF endpoint among Week 1 - 6; n= 128, 126, 128; number of subjects who responded to the scale.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
score on scale | -5.78 (1.01) | -5.43 (1.02) | -6.79 (1.02)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.3299, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.1915, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]

15. Secondary Outcome: Change in Quality of Life, Enjoyment, and Satisfaction Scale (Q-LES-Q) Total Score at Endpoint
Description: Change is observed value at each visit minus baseline value. LOCF endpoint among Week 1 through Week 6. Q-LES-Q: 16-item instrument for patients assessment of his/her quality of life; overall level of satisfaction scale 1=very poor to 5=Very good (1 item re medication can be blank). Total possible score 15 - 80
Time Frame: Baseline to 6 Weeks
Population: ITT Population Observed Cases.n= 142, 137, 139; number of subjects who responded to the scale. Endpoint is LOCF endpoint among Week 1 through Week 6.
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
score on scale | 0.08 (0.02) | 0.09 (0.02) | 0.09 (0.02)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.5407, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.6079, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]

16. Secondary Outcome: Change in Bech Melancholia Score
Description: Change is observed value at each visit minus baseline value. Endpoint is LOCF endpoint among Week 1 through Week 6. Bech Melancholia is the sum of Scores on 6 Items pertaining to melancholia within Hamilton Depression Rating Scale (HAM-D). Scale 0 to 4, higher scores reflecting greater severity;Total possible 0 - 24.
Time Frame: Baseline to 6 Weeks
Population: ITT Population Observed cases
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
score on scale
  Week 3 (n = 147, 149, 148) | -5.12 (0.47) | -5.61 (0.47) | -5.22 (0.47)
  Week 6 (n = 104, 117, 125) | -6.91 (0.65) | -6.93 (0.62) | -6.23 (0.61)
  Endpoint (n =151, 150, 153) | -5.85 (0.54) | -6.23 (0.54) | -5.70 (0.54)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.8464, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.4023, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: 120-160mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.2870, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.2537, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.7909, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.3308, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]

17. Secondary Outcome: Change in Anxiety/Somatizations Factor Total Score
Description: Change is observed value at each visit minus baseline value. Endpoint is LOCF endpoint among Week 1 through Week 6. This instrument = sum of Scores on 6 Items measuring anxiety/somatization within Hamilton Depression Rating Scale (HAM-D). Scale range is 0 to 4, higher scores reflecting greater severity. Total possible 0 - 24.
Time Frame: Baseline to 6 Weeks
Population: ITT Population Observed Cases
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
score on scale
  Week 3 (n = 147,149,148) | -2.69 (0.30) | -2.92 (0.30) | -2.98 (0.30)
  Week 6 (n = 104,117,125) | -3.67 (0.40) | -3.88 (0.38) | -3.62 (0.38)
  Endpoint (n = 151,150,153) | -3.04 (0.34) | -3.39 (0.34) | -3.32 (0.34)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.3355, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.8447, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: 120-160mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.8959, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.4826, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.4178, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.8277, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 4, analysis 1]

18. Secondary Outcome: Change in Retardation Factor Scores
Description: Change is observed value at each visit minus baseline value. This instrument = sum of Scores of 4 items on retardation within Hamilton Depression Rating Scale (HAM-D). Scale range is 0 to 4 with higher scores reflecting greater severity. Total possible is 0 - 16.
Time Frame: Baseline to 6 Weeks
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
score on scale
  Week 3 (n = 147,149,148) | -3.50 (0.32) | -3.64 (0.32) | -3.59 (0.33)
  Week 6 (n = 104,117,125) | -4.44 (0.42) | -4.40 (0.40) | -3.79 (0.40)
  Endpoint (n = 151,150,153) | -3.89 (0.35) | -3.99 (0.35) | -3.62 (0.35)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.7758, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.8737, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: 120-160mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.1151, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.1290, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.4432, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.2988, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]

19. Secondary Outcome: Change in Sleep Disturbance Factor Score
Description: Change is observed value at each visit minus baseline value. Endpoint is LOCF endpoint among Week 1 through Week 6. This instrument = sum of Scores of 3 items on sleep disturbance within Hamilton Depression Rating Scale (HAM-D). Scale range 0 to 4 with higher scores reflecting greater severity. Total possible is 0 - 12.
Time Frame: Baseline to 6 weeks
Population: ITT Population Observed cases
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
score on scale
  Week 3 (n = 147, 149, 148) | -1.92 (0.24) | -2.07 (0.23) | -1.96 (0.24)
  Week 6 (n = 104, 117, 125) | -2.20 (0.30) | -2.19 (0.28) | -2.06 (0.28)
  Endpoint (n = 151, 150 153) | -1.90 (0.24) | -1.98 (0.24) | -1.96 (0.24)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.8598, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 3; Test type: Superiority or Other; p = 0.6513, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: 120-160mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.6272, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: 40-80 mg Ziprasidone vs Placebo; Week 6; Test type: Superiority or Other; p = 0.6467, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.8049, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.9411, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]

20. Secondary Outcome: Change in Verbal Memory Trial Performance Total Score at Endpoint
Description: Change is observed value at each visit minus baseline value. Endpoint is LOCF endpoint among Week 1 through Week 6. This test is part of Brief Assessment of Cognition and measures recall of 15 words repeated 5 times. Range 0-75 words, higher number reflects better recall.
Time Frame: Baseline to 6 Weeks LOCF
Population: Intent to Treat (ITT) population observed cases. Endpoint is LOCF endpoint among Week 1 through Week 6.
Measure: Least Squares Mean (Standard Error); unit: words
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
words | 1.31 (0.97) | 0.85 (0.96) | 1.22 (1.00)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.9260, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.7100, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]

21. Secondary Outcome: Change in Affective Interference Test Immediate Recall List 1 Emotional Words at Endpoint
Description: Change is observed value at each visit minus baseline value. Endpoint is LOCF endpoint among Week 1 through Week 6. This is a test in Brief Assessment of Cognition measuring immediate recall of 15 emotional words; higher number of words is better recall.
Time Frame: Baseline to 6 Weeks LOCF
Population: Intent to treat (ITT) population observed cases
Measure: Least Squares Mean (Standard Error); unit: words
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
words | -0.28 (0.15) | -0.30 (0.15) | -0.06 (0.16)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.1836, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.1374, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]

22. Secondary Outcome: Change in Affective Interference Test Immediate Recall Non-Emotional Words List 1 at Endpoint
Description: Change is observed value at each visit minus baseline value. Endpoint is LOCF endpoint among Week 1 through Week 6. This instrument measures immediate recall of 15 non-emotional words (List 1); higher number of words is better recall.
Time Frame: Baseline to 6 Weeks LOCF
Population: Intent to treat (ITT) population observed cases
Measure: Least Squares Mean (Standard Error); unit: words
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
words | -0.02 (0.15) | 0.14 (0.15) | -0.00 (0.16)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.9237, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.3786, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]

23. Secondary Outcome: Change in Affective Interference Test, Immediate Recall, List 2 Emotional Words at Endpoint
Description: Change is observed value at each visit minus baseline value. Endpoint is LOCF endpoint among Week 1 through Week 6. This test is in Brief Assessment of Cognition and measures immediate recall of 15 emotional words (List 2); higher number of words is better recall
Time Frame: Baseline to 6 Weeks LOCF
Population: Intent to treat (ITT) population observed cases. Endpoint is LOCF endpoint among Week 1 through Week 6.
Measure: Least Squares Mean (Standard Error); unit: words
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
words | -0.09 (0.19) | -0.05 (0.19) | 0.05 (0.19)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.4624, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.5971, ANCOVA; [statistical method as in outcome 4, analysis 1]

24. Secondary Outcome: Change in Affective Interference Test, Immediate Recall, List 2 Non-Emotional Words at Endpoint
Description: Change is observed value at each visit minus baseline value. Endpoint is LOCF endpoint among Week 1 through Week 6. This is a test in Brief Assessment of Cognition which measures immediate recall of 15 non-emotional words (List 2); higher number of words is better recall
Time Frame: Baseline to 6 Weeks LOCF
Population: Intent to treat (ITT) population observed cases. Endpoint is LOCF endpoint among Week 1 through Week 6.
Measure: Least Squares Mean (Standard Error); unit: words
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
words | -0.16 (0.19) | 0.07 (0.19) | 0.13 (0.20)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.1378, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.7665, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]

25. Secondary Outcome: Change in Affective Interference Test, Immediate Recall, List 3 Emotional Words at Endpoint
Description: Change is observed value at each visit minus baseline value. Endpoint is LOCF endpoint among Week 1 through Week 6. This is a test in Brief Assessment of Cognition which measures immediate recall of 15 emotional words (List 3); higher number of words is better recall
Time Frame: Baseline to Week 6 LOCF
Population: Intent to treat (ITT) population observed cases.Endpoint is LOCF endpoint among Week 1 through Week 6.
Measure: Least Squares Mean (Standard Error); unit: words
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
words | -0.18 (0.21) | -0.30 (0.20) | -0.03 (0.21)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.4767, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.2066, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]

26. Secondary Outcome: Change in Affective Interference Test, Immediate Recall, List 3 Non-Emotional Words at Endpoint
Description: Change is observed value at each visit minus baseline value. Endpoint is LOCF endpoint among Week 1 through Week 6. This is a test in Brief Assessment of Cognition which measures immediate recall of 15 non-emotional words (List 3); higher number of words is better recall
Time Frame: Baseline to Week 6 LOCF
Population: Intent to treat (ITT) population observed cases
Measure: Least Squares Mean (Standard Error); unit: words
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
words | -0.52 (0.19) | -0.15 (0.19) | -0.24 (0.20)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.1667, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.6727, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]

27. Secondary Outcome: Change in Affective Interference Test, Immediate Recall, Cued-Recall Non-Emotional Words at Endpoint
Description: Change is observed value at each visit minus baseline value. Endpoint is LOCF endpoint among Week 1 through Week 6. This is a test in Brief Assessment of Cognition which measures immediate recall (Cued) of 15 non-emotional words; higher number of words is better recall
Time Frame: Baseline to 6 Weeks LOCF
Population: Intent to treat (ITT) population observed cases. Endpoint is LOCF endpoint among Week 1 through Week 6.
Measure: Least Squares Mean (Standard Error); unit: words
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
words | -0.39 (0.18) | -0.01 (0.18) | -0.32 (0.19)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.7019, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.1020, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]

28. Secondary Outcome: Change in Affective Interference Test, Immediate Recall, Cued-Recall Emotional Words at Endpoint
Description: Change is observed value at each visit minus baseline value. Endpoint is LOCF endpoint among Week 1 through Week 6. This is a test in Brief Assessment of Cognition which measures immediate recall (Cued) of 15 emotional words; higher number of words is better recall
Time Frame: Baseline to 6 Weeks LOCF
Population: Intent to treat (ITT) population observed cases. Endpoint is LOCF endpoint among Week 1 through Week 6.
Measure: Least Squares Mean (Standard Error); unit: words
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
words | -0.06 (0.20) | -0.07 (0.20) | 0.08 (0.20)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.4749, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.4491, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]

29. Secondary Outcome: Change in Digit Sequencing Task at Endpoint
Description: Change is observed value at each visit minus baseline value. Endpoint is LOCF endpoint among Week 1 through Week 6. This is a test in Brief Assessment of Cognition in which patient sequences digits from lowest to highest. Range of number of correct responses (0-28); higher numbers show better digit sequencing and greater cognition.
Time Frame: Baseline to 6 Weeks LOCF
Population: Intent to treat (ITT) population observed cases
Measure: Least Squares Mean (Standard Error); unit: Number Correct
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
Number Correct | 0.76 (0.37) | 0.09 (0.37) | 0.46 (0.38)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.4398, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.3331, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 4, analysis 1]

30. Secondary Outcome: Change in Token Motor Task at Endpoint
Description: Change is observed value at each visit minus baseline value. Endpoint is LOCF endpoint among Week 1 through Week 6. This is a test in Brief Assessment of Cognition in which a patient places as many of 100 tokens (2 at a time) into a container as they can within 60 seconds. The higher number of tokens placed = patient is better at motor tasks
Time Frame: Baseline to 6 Weeks LOCF
Population: Intent to treat (ITT) population observed cases. Endpoint is LOCF endpoint among Week 1 through Week 6.
Measure: Least Squares Mean (Standard Error); unit: Number of Tokens
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
Number of Tokens | 0.28 (1.54) | -0.00 (1.53) | 2.02 (1.57)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.2763, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.2048, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 4, analysis 1]

31. Secondary Outcome: Change in Verbal Fluency in Naming Categories at Endpoint
Description: Change is observed value at each visit minus baseline value. Endpoint is LOCF endpoint among Week 1 through Week 6. This is a test in Brief Assessment of Cognition.Patients are given 60 seconds to name as many words as possible within a given category. The more words named=better cognition.
Time Frame: Baseline to 6 Weeks LOCF
Population: Intent to treat (ITT) population observed cases.Endpoint is LOCF endpoint among Week 1 through Week 6.
Measure: Least Squares Mean (Standard Error); unit: Number Correct
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
Number Correct | 0.19 (0.58) | -0.11 (0.58) | -0.28 (0.60)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.4340, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.7774, ANCOVA — For all efficacy analyses, no multiple comparisons adjustments were made; [statistical method as in outcome 4, analysis 1]

32. Secondary Outcome: Change in Verbal Fluency Controlled Word Association at Endpoint
Description: Change is observed value at each visit minus baseline value. Endpoint is LOCF endpoint among Week 1 through Week 6. This is a test in Brief Assessment of Cognition. Patients given 60 seconds to generate as many words as possible that begin with a given letter; better verbal fluency = more words
Time Frame: Baseline to 6 Weeks LOCF
Population: Intent to treat (ITT) population observed cases. Endpoint is LOCF endpoint among Week 1 through Week 6.
Measure: Least Squares Mean (Standard Error); unit: Number Correct
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
Number Correct | 1.09 (0.67) | -0.15 (0.66) | 1.54 (0.69)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.5195, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.0153, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]

33. Secondary Outcome: Change in Symbol Coding at Endpoint
Description: Change is observed value at each visit minus baseline value. Endpoint is LOCF endpoint among Week 1 through Week 6. This is a test in Brief Assessment of Cognition. For 90 seconds, Patient writes numerals 1-9 as matched to symbols. Range 0 to 110 with higher totals = better cognition.
Time Frame: Baseline to 6 Weeks LOCF
Population: Intent to treat (ITT) population observed cases. Endpoint is LOCF endpoint among Week 1 through Week 6.
Measure: Least Squares Mean (Standard Error); unit: Total Correct
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
Total Correct | 1.34 (1.18) | 1.07 (1.16) | 2.66 (1.21)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.2847, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.1958, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]

34. Secondary Outcome: Change in Tower of London Test at Endpoint
Description: Change is observed value at each visit minus baseline value. Endpoint: LOCF endpoint among Week 1 through Week 6. Brief Assessment of Cognition: subjects asked to arrange balls in 2 pictures so they are identical and give the total number of ball movements to reach this arrangment. Range: 0-22; more correct = better cognition.
Time Frame: Baseline to 6 Weeks LOCF
Population: Intent to treat (ITT) population observed cases. Endpoint is LOCF endpoint among Week 1 through Week 6.
Measure: Least Squares Mean (Standard Error); unit: Number Correct
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
Number Correct | 0.31 (0.41) | 0.68 (0.41) | 0.91 (0.43)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.1652, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.5997, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]

35. Secondary Outcome: Change in Affective Interference Test, Delayed Recognition, Emotional Words at Endpoint
Description: Change is observed value at each visit minus baseline value. Endpoint is LOCF endpoint among Week 1 through Week 6. Test in Brief Assessment of Cognition in which the number of correct emotional words in delayed recognition is measured. Range 0-75 with higher numbers showing better cognition.
Time Frame: Baseline to 6 Weeks LOCF
Population: Intent to treat (ITT) population observed cases. Endpoint is LOCF endpoint among Week 1 through Week 6
Measure: Least Squares Mean (Standard Error); unit: Words
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
Words | -0.37 (0.22) | 0.15 (0.22) | 0.23 (0.22)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.0082, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.7037, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]

36. Secondary Outcome: Change in Affective Interference Test, Delayed Recognition, Emotional Words False Alarms at Endpoint
Description: Change is observed value at each visit minus baseline value. Endpoint is LOCF endpoint among Week 1 through Week 6. Test in Brief Assessment of Cognition which measures number of correct emotional word's false alarms (during delayed recognition). Higher number = better cognition
Time Frame: Baseline to 6 Weeks LOCF
Population: Intent to treat (ITT) population observed cases. Endpoint is LOCF endpoint among Week 1 through Week 6.
Measure: Least Squares Mean (Standard Error); unit: Number Correct
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
Number Correct | 0.09 (0.10) | 0.01 (0.10) | -0.03 (0.10)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.2718, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.7077, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]

37. Secondary Outcome: Change in Affective Interference Test, Delayed Recognition, Non-Emotional Words at Endpoint
Description: Change is observed value at each visit minus baseline value. Endpoint is LOCF endpoint among Week 1 through Week 6. This is a test in Brief Assessment of Cognition which measures number of Non-Emotional Words (Delayed Recognition); higher number of words = better cognition
Time Frame: Baseline to Week 6 LOCF
Population: Intent to treat (ITT) population observed cases. Endpoint is LOCF endpoint among Week 1 through Week 6.
Measure: Least Squares Mean (Standard Error); unit: Number Correct
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
Number Correct | -0.18 (0.23) | -0.24 (0.23) | -0.02 (0.24)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.5057, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.3654, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]

38. Secondary Outcome: Change in Affective Interference Test, Delayed Recognition, Non-Emotional Words False Alarms at Endpoint
Description: Change is observed value at each visit minus baseline value. Endpoint is LOCF endpoint among Week 1 through Week 6. This is a test in Brief Assessment of Cognition which measures number of correct non-eEmotional word's false alarms(at delayed recognition). Higher number of words = greater cognition
Time Frame: Baseline to Week 6 LOCF
Population: Intent to treat (ITT) population observed cases. Endpoint is LOCF endpoint among Week 1 through Week 6.
Measure: Least Squares Mean (Standard Error); unit: Number Correct
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Number analyzed (Participants) | 166 | 158 | 162
Number Correct | 0.06 (0.15) | 0.19 (0.15) | 0.14 (0.16)
Statistical Analysis 1: Comparison: 120-160mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.6227, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: 40-80 mg Ziprasidone vs Placebo; Endpoint; Test type: Superiority or Other; p = 0.7737, ANCOVA — For all secondary efficacy analyses, no multiple comparison adjustment were made; [statistical method as in outcome 4, analysis 1]

ADVERSE EVENTS:
Arm/Group | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Serious Adverse Events (participants affected / at risk) | 7 | 3 | 6
Other Adverse Events (participants affected / at risk) | 89 | 70 | 57
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Abdominal pain (Gastrointestinal disorders) | 1/171 | 0/165 | 0/168
Oedema peripheral (General disorders) | 1/171 | 0/165 | 0/168
Pneumonia (Infections and infestations) | 0/171 | 1/165 | 0/168
Upper respiratory tract infection (Infections and infestations) | 1/171 | 0/165 | 0/168
Urinary tract infection (Infections and infestations) | 1/171 | 1/165 | 0/168
Road traffic accident (Injury, poisoning and procedural complications) | 0/171 | 1/165 | 0/168
Back pain (Musculoskeletal and connective tissue disorders) | 0/171 | 1/165 | 0/168
Bipolar I disorder (Psychiatric disorders) | 1/171 | 0/165 | 1/168
Depression (Psychiatric disorders) | 0/171 | 1/165 | 1/168
Depression suicidal (Psychiatric disorders) | 1/171 | 0/165 | 1/168
Hallucination, auditory (Psychiatric disorders) | 0/171 | 1/165 | 0/168
Mania (Psychiatric disorders) | 0/171 | 0/165 | 1/168
Psychotic disorder (Psychiatric disorders) | 0/171 | 0/165 | 1/168
Suicidal ideation (Psychiatric disorders) | 0/171 | 1/165 | 1/168
Nephrolithiasis (Renal and urinary disorders) | 1/171 | 0/165 | 0/168
Rash (Skin and subcutaneous tissue disorders) | 1/171 | 0/165 | 0/168
Swelling face (Skin and subcutaneous tissue disorders) | 1/171 | 0/165 | 0/168
Hypertension (Vascular disorders) | 1/171 | 0/165 | 0/168
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | 120-160mg Ziprasidone | 40-80 mg Ziprasidone | Placebo
Diarrhoea (Gastrointestinal disorders) | 2/171 | 8/165 | 14/168
Dry mouth (Gastrointestinal disorders) | 13/171 | 6/165 | 5/168
Nausea (Gastrointestinal disorders) | 17/171 | 10/165 | 11/168
Dizziness (Nervous system disorders) | 12/171 | 6/165 | 7/168
Headache (Nervous system disorders) | 16/171 | 18/165 | 13/168
Sedation (Nervous system disorders) | 20/171 | 8/165 | 2/168
Somnolence (Nervous system disorders) | 30/171 | 25/165 | 8/168
Anxiety (Psychiatric disorders) | 9/171 | 3/165 | 5/168
Insomnia (Psychiatric disorders) | 16/171 | 9/165 | 8/168

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 mo from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.